CLINICAL TRIAL: NCT00139490
Title: Home-Based Blood Pressure Interventions for African Americans
Brief Title: Home-Based Program to Treat High Blood Pressure in African Americans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Visiting Nurse Service of New York (Other)
Responsible Party: Penny Feldman, PhD, Principal Investigator, Visiting Nurse Service of New York
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 246; R01HL078585 (NIH)
Record Dates: First submitted 2005-08-29; First posted 2005-08-31 (Estimated); Last update posted 2012-12-21 (Estimated); Status verified 2012-12

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension
Keywords: Blood Pressure, High
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A (Experimental): The augmented intervention will consist of just-in-time nurse, patient and physician information and feedback during the post-acute period, plus transition to an ongoing Home-Based HTN Support Program within approximately 30 days after the patient's admission to home health care. The augmented intervention adds an HTN Nurse Specialist (advanced practice nurse) and a lay community health worker, who will be responsible for assuring a patient's smooth transition to the Home-Based HTN Support Program and for delivering the main components of that intervention, backed up by the project physician.
  Interventions: Behavioral: Health Education Program
- B (Active Comparator): The basic information and referral intervention will deliver key "just-in-time" information to nurses, patients and patients' physicians while the patient is receiving post-acute home care services. The basic intervention relies on care provided by home health nurses during the routine home health stay.
  Interventions: Behavioral: Basic Group
- C (Placebo Comparator): Usual Care group
  Interventions: Behavioral: Control Group

INTERVENTIONS:
Behavioral: Health Education Program — The augmented intervention will consist of just-in-time nurse, patient and physician information and feedback during the post-acute period, plus transition to an ongoing Home-Based HTN Support Program within approximately 30 days after the patient's admission to home health care. The augmented intervention adds an HTN Nurse Specialist (advanced practice nurse) and a lay community health worker, who will be responsible for assuring a patient's smooth transition to the Home-Based HTN Support Program and for delivering the main components of that intervention, backed up by the project physician.
  Arms: A
Behavioral: Basic Group — The basic information and referral intervention will deliver key "just-in-time" information to nurses, patients and patients' physicians while the patient is receiving post-acute home care services. The basic intervention relies on care provided by home health nurses during the routine home health stay.
  Arms: B
Behavioral: Control Group — Usual Care
  Arms: C

SUMMARY:
The purpose of this study is to examine the effectiveness and cost effectiveness of two organizational interventions aimed at improving blood pressure (BP) control among a high-risk, African American home care population.

DETAILED DESCRIPTION:
BACKGROUND:

Home health care is a non-institutional, "diverse health care setting" that provides services to a high-risk population characterized by multiple chronic conditions and significant needs for both medical and self-care management. Home health agencies discharged approximately 7.6 million patients in 1998, of whom approximately 60 to 65% were female and 12 to 15% black (US DHHS 2000; Haupt 1998). Home health patients are clinically diverse. Individuals with conditions of the circulatory system comprise the single largest share (about 22% in 1996) (Haupt 1998), while heart failure (I-IF), diabetes, chronic obstructive pulmonary disease, and essential hypertension (HTN) are patients' most frequent primary diagnoses (Haupt & Jones 1999). Most home health patients enter care after a hospitalization and more than two-thirds are discharged to the community. Management of HTN has not been a high priority for guideline adoption or quality improvement activities in home health care (Peterson 2004), even though approximately 8% of home care patients are admitted with essential HTN as a first, second, or third diagnosis (Haupt & Jones, 1999). In the words of one clinical nurse specialist, home health nurses tend to see elevated BP readings as "a set of numbers rather than a condition to be managed," despite the fact that their patients may be at high risk of future HTN-related complications by virtue of their comorbidities and history of prior hospitalization.

Teaching patients about their conditions, promoting patient self-management, helping patients adhere to medical regimens established by their physicians, and linking them to community resources are central to the role of the home health nurse (Clemen-Stone et al. 2002). However, with the advent of a home health prospective payment system, nurses are working under heightened pressure to constrain service use and reduce time in the patient's home. This pressure, in turn, may provide a disincentive to focus on high BP management issues, particularly when HTN is a second or third diagnosis and not the primary reason for which a person has been admitted to home care. Thus home health care represents a segment of the health care system where a significant number of high-risk HTN patients are served, where HTN practice likely requires significant improvement, and where nursing personnel are uniquely positioned to mobilize their care management and patient education skills to increase the proportion of treated HTN patients who achieve adequate BP control. The underlying premise of the project is that organizational change to improve BP management and outcomes will not easily occur in home health care without new intervention models, rigorous evaluation of their impact, or efforts by opinion leaders in the clinical and research communities to disseminate information on strategies that are efficacious and cost-effective. Visiting Nurse Service of New York (VNSNY), serving over 70,000 adult patients per year, provides a prominent organizational "laboratory" for testing promising new models of care.

The study is in response to a Request for Applications released in September 2003 on "Interventions to Improve Hypertension Control Rates in African Americans."

DESIGN NARRATIVE:

The study will enroll African American patients with uncontrolled hypertension who are entering the home care program of the VNSNY. It will employ a randomized design, whereby all VNSNY nurses who are providing direct care to the eligible study population (an estimated 300 nurses serving an estimated 1000 African American patients with uncontrolled hypertension) will be randomly assigned to a control group or one of two intervention groups upon identification of the first eligible hypertensive patient to whom they provide care during the study period. Throughout the study, each nurse will continue to administer the same intervention, either usual care, basic intervention, or an augmented intervention, so that randomization will be by nurse, rather than by patient. A nurse's initial random assignment to a specific group (usual care, basic treatment, or augmented treatment) will determine the status for all new patients allocated to that particular nurse's care for the duration of the study.

The two interventions to be tested include the following: 1) a "basic" intervention delivering key evidence-based information to nurses, physicians, and patients while the patient is receiving traditional post-acute home health care; and 2) an "augmented" intervention transitioning patients to a Home-Based HTN Support Program that extends the information, monitoring, and feedback available to patients and primary care physicians for a 12-month period beyond an index home care admission. The interventions will be assessed relative to usual care and to each other. The analysis will estimate the impact of the basic and augmented interventions on nursing practices and processes of care, patient hypertension management (e.g., medication adherence), BP outcomes, and overall costs. Behaviors and outcomes will be measured at fixed points in time. Measures will be derived from a combination of primary and secondary data, including patient records, patient assessment instruments, patient interviews, home BP monitors, urine tests, and administrative files. Multivariate regression analyses will be conducted to determine intervention effects on study outcomes, adjusting for selected nurse and patient characteristics. Nurse level risk-adjustment will include demographics and other measures that might influence practice or processes of care, such as experience and education. Patient-level risk adjustment will include demographics, social support, and other characteristics that might influence behavior, service use, BP, or other health outcomes. Estimates of treatment-control group differences (for both treatments) generated by these models will be tested to determine the extent to which observed differences at the nurse and patient levels are attributable to the alternative intervention strategies.

ELIGIBILITY:
Inclusion Criteria:

* African American
* Have uncontrolled hypertension, defined as BP greater than 140/90 mm Hg (systolic, diastolic, or both), and 130/80 mm Hg for individuals with diabetes or kidney failure

Exclusion Criteria:

* Severe heart failure
* Moderate to severe cognitive impairment
* Overall "poor" or "guarded" prognosis
* Life expectancy of less than 6 months from study entry

Ages: 21 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 846 (Actual)
Dates: Start 2006-02; Primary Completion 2009-05 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Documented adherence to nursing-specific practices that reflect and reinforce JNC7 guidelines | Measured at 12 months
Change in systolic and diastolic BP | Measured at 12 months
Proportion of patients that are below the target home BP levels (135/85 mm Hg for non-diabetic and kidney disease participants; 125/75 mm Hg for diabetic and kidney disease participants | Measured at 12 months
Changes in systolic and diastolic Blood Pressure | Measured at 12 months

SECONDARY OUTCOMES:
Medication adherence | Measured at 12 months
Sodium intake | Measured at 12 months
Health care utilization | Measured at 12 months
Cost-effectiveness of the program | Measured at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Penny H. Feldman, PhD, Principal Investigator — Center for Home Care Policy & Research, Visiting Nurse Service of New York

REFERENCES:
- [Derived] Feldman PH, McDonald MV, Barron Y, Gerber LM, Peng TR. Home-based interventions for black patients with uncontrolled hypertension: a cluster randomized controlled trial. J Comp Eff Res. 2016 Mar;5(2):155-68. doi: 10.2217/cer.15.60. Epub 2016 Mar 7. PMID 26946952